CLINICAL TRIAL: NCT02739841
Title: Acute Hemodynamic Responses to Ventilator Hyperinflation Technique in Critical Traumatic Patients With Pulmonary Complications
Brief Title: Hemodynamic Responses to Ventilator Hyperinflation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Mr.Atsadang Natisri, Principal Investigator, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VHI-hemodynamic responses
Record Dates: First submitted 2016-01-28; First posted 2016-04-15 (Estimated); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Complications
Keywords: hemodynamic response

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ventilator hyperinflation (Experimental): For the ventilator hyperinflation techniques (VHI), the study consists of three consecutive periods 1) baseline period: 10 minutes rest in side lying by effected lung uppermost with head-up 30 degree 2) Intervention period: Patients were positioned as same as baseline period and 4 sets of 6 hyperinflation breath were applied by mechanical ventilator at 150% of tidal volume (VT) at initial 3) recovery period: 10 minutes rest in the same position but reduce VT to initial.
  Interventions: Other: Ventilator hyperinflation
- Chest physical therapy (Experimental): For the conventional chest physical therapy (CPT), the study will be performed in the similar procedure except the intervention period, the patient will be received vibration and passive of the both upper extremity.
  Interventions: Other: Chest physical therapy

INTERVENTIONS:
Other: Ventilator hyperinflation — 4 sets of 6 hyperinflation breath were applied by mechanical ventilator at 150% of tidal volume (VT) at initial.
  Arms: Ventilator hyperinflation
Other: Chest physical therapy — The patient will be received vibration and passive of the both upper extremity.
  Arms: Chest physical therapy

SUMMARY:
The purpose of this study is to explore acute hemodynamic responses to VHI technique in critical traumatic patients with pulmonary complications in the intensive care unit.

DETAILED DESCRIPTION:
The World Health Organization reported that Thailand ranked third for number of road fatalities at 38.1 per 100,000 inhabitants in 2010. Most of these cases were admitted to the intensive care unit (ICU) for respiratory interventions such as intubation and mechanical ventilation that can lead to a common problem of pulmonary complications such as pneumonia and atelectasis.

Evidence supports the effectiveness of chest physical therapy technique (CPT) to improve alveolar collapse and remove pulmonary secretion. A previous study has shown that the positive airway pressure technique reduced work of breathing (WOB) and re-inflated lung atelectasis. The use of positive pressure devices has been part of physiotherapy intervention since intermittent positive pressure breathing was introduced in clinical practice. In intensive care settings, the use of positive pressure by physiotherapists includes manual hyperinflation (bagging or bag squeezing), which has been shown to increase oxygenation and mobilize excessive bronchial secretions, and to re-inflate collapsed areas.

Manual hyperinflation technique (MHI) is provided for use in patients with lung atelectasis. Several studies demonstrated the short-term effects of increased oxygenation and pulmonary compliance, improved lung collapse, and removed pulmonary secretions. To apply MHI technique, patients were disconnected from the ventilator which lead to the adverse effect of losing positive end expiratory pressure (PEEP) corresponding to loss of functional residual capacity, decreased oxygenation, and shear stress of distal lung units.

An alternative method of performing pulmonary hyperinflation uses the mechanical ventilator. Although there is evidence that positive pressure interventions such as continuous positive airway pressure (CPAP) and intermittent positive pressure breathing IPPB) can improve lung expansion and mobilize secretions in the airway, there are few studies examining ventilator-induced hyperinflation as a physiotherapy intervention in intensive care.

A previous study showed that the ventilator hyperinflation technique (VHI) was as effective as MHI to improve pulmonary complications such as secretion retention and lung atelectasis. Especially, VHI technique using applied by the mechanical ventilator, patient was not disconnected from the ventilator and therefore did not result in loss of PEEP and its adverse effect.

Atelectasis is a common pulmonary complication in acute trauma patients maintained on ventilator support who would benefit from VHI but even though recent studies indicate that VHI technique is an improvement on the MHI technique there are relatively few study of the hemodynamic responses to VHI. There is controversy in hemodynamic responses to VHI, Ventilator hyperinflation technique (VHI) is especially valuable in treating patients in the ICU because other techniques such as percussion and postural drainage may not be possible because of wounds, broken bones or surgical drains. However, the technique is very rarely used by physical therapists in the ICU, possibly because they are concerned that increasing in the intra-thoracic pressure by uses VHI to inflate lung will result in dangerous changes in heart rate and blood pressure; that any such changes may persist after the treatment leading to complications such as pulmonary edema and, lastly, the positive pressure to the patient may precipitate episodes of cardiac arrhythmia.

Recent study demonstrated that heart rate and blood pressure were changed after VHI in ICU patients but the condition of patients in their study were mixed, not only traumatic patients. Previous study showed that basal heart and blood pressure were increased in patients underwent traumatic conditions. The hemodynamic responses to VHI were required for safety and increasing physiotherapist's confidences to use this technique in ICU. Therefore, the purpose of this study is to explore acute hemodynamic responses to VHI technique in critical traumatic patients with pulmonary complications in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanical ventilator dependence

Exclusion Criteria:

1. acute respiratory distress syndrome (ARDS)
2. acute lung injury (ALI)
3. pulmonary contusion
4. undrained pneumothorax, hemothoarax, and hemopneumothorax
5. bronchospasm
6. pulmonary bullae/blebs
7. lung tumors
8. lung abscess
9. haemoptysis
10. mean arterial pressure (MAP) <70 mmHg
11. positive end expiratory pressure (PEEP) >6 cm H2O
12. heart rate (HR) > 140 beats/min
13. blood pressure (BP) <90/60 or >180/100 mmHg
14. restlessness
15. oxygen saturation (SpO2) < 90 %
16. spontaneous respiratory rate (RR) > 35 beats/min

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure (MAP) | "change from baseline in mean arterial pressure (MAP) at during intervention" and "change from baseline in mean arterial pressure (MAP) at immediately after intervention"
  Change from baseline in mean arterial pressure (MAP)

SECONDARY OUTCOMES:
Heart rate (HR) | "change from baseline in heart rate (HR) at during intervention" and "change from baseline in heart rate (HR) at immediately after intervention"
  Change from baseline in heart rate (HR)
Systolic blood pressure (SBP) | "change from baseline in systolic blood pressure (SBP) at during intervention" and "change from baseline in systolic blood pressure (SBP) at immediately after intervention"
  Change from baseline in systolic blood pressure (SBP)
Diastolic blood pressure (DBP) | "change from baseline in diastolic blood pressure (DBP) at during intervention" and "change from baseline in diastolic blood pressure (DBP) at immediately after intervention"
  Change from baseline in diastolic blood pressure (DBP)
Central venous pressure (CVP) | "change from baseline in central venous pressure (CVP) at during intervention" and "change from baseline in central venous pressure (CVP) at immediately after intervention"
  Change from baseline in central venous pressure (CVP)

CONTACTS AND LOCATIONS:
Overall Officials: Atsadang Natisri, Master, Principal Investigator — school of physical therapy, faculty of associated medical sciences
Locations (1):
- School of physical therapy, Faculty of Associated Medical Science, Khon Kaen University, Khon Kaen, Thailand